CLINICAL TRIAL: NCT04460729
Title: A Phase II, Open-Label, Multicenter Study of Capmatinib in Subjects With MET Exon 14 Skipping Mutation Positive, Advanced, Non Small-Cell Lung Cancer That Has Metastasized to the Brain
Brief Title: A Phase II, Open-Label, Multicenter Study of Capmatinib in Subjects With MET Exon 14 Skipping Mutation Positive, Advanced, NSCLC With Brain Metastases
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: company decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CINC280A2203
Record Dates: First submitted 2020-07-02; First posted 2020-07-08 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Non-small Cell Lung Carcinoma (NSCLC)
Keywords: Non-small cell lung carcinoma; Non-small cell lung cancer; NSCLC; Treatment of lung cancer after first metastasi; Lung cancer; Lung adenocarcinoma; Squamous cell lung carcinoma; Large-cell lung carcinoma; Large-cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Adenocarcinoma of Lung | interventions — capmatinib

STUDY DESIGN:
Intervention Model Description: Approximately 60 participants will be enrolled globally and allocated to one of two cohorts based on whether their metastatic brain disease is symptomatic or asymptomatic and with or without prior brain therapy or if they have been diagnosed with leptomeningeal disease
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Participants who are asymptomatic and without prior brain therapy
  Interventions: Drug: Capmatinib
- Cohort 2 (Experimental): Participants who are symptomatic with or without prior brain therapy or asymptomatic with prior brain therapy or with leptomeningeal disease
  Interventions: Drug: Capmatinib

INTERVENTIONS:
Drug: Capmatinib — 400 mg administered orally twice daily

SUMMARY:
The purpose of this study is to establish the intracranial efficacy of single agent capmatinib in the population of treatment-naïve or pretreated with one or two prior lines of systemic therapies for advanced stage Non Small-Cell Lung Cancer (NSCLC) with MET exon 14 mutation that has metastasized to the brain.

Cohort 1 (asymptomatic brain metastases (BM) without prior brain therapy) has been selected to identify patients who are most likely to benefit from capmatinib therapy in this setting and to establish a clinically relevant response outcome.

Cohort 2 is a heterogeneous group of patients (symptomatic with and without prior brain therapy, asymptomatic with prior brain therapy, or with leptomeningeal disease.), and the outcomes will be descriptive only

DETAILED DESCRIPTION:
This is a prospectively designed, multicenter, open-label, two-cohort, phase II study to evaluate the intracranial efficacy of single agent capmatinib in participants with MET exon 14 mutated NSCLC and BM. Participants can be treatment naïve or pretreated with one or two prior lines of systemic therapies for advanced stage (stage IIIb - IV) NSCLC.

Approximately 60 participants will be enrolled globally and allocated to one of two cohorts:

Cohort 1 will enroll approximately 40 participants who are asymptomatic and without prior brain therapy.

Cohort 2 will enroll approximately 20 participants who are symptomatic with or without prior brain therapy or asymptomatic with prior brain therapy or with leptomeningeal disease.

All participants will be pre-screened for MET mutation and presence of BM will be documented at baseline by a radiologist/neuroradiologist.

Intracranial disease will be assessed and response to treatment will be evaluated using the Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM) criteria every 8 weeks. Extracranial and whole body disease will be assessed and response to treatment will be evaluated using RECIST 1.1 every 8 weeks.

Participants will receive capmatinib 400 mg b.i.d. until they experience any of the following: documented disease progression by RANO-BM criteria and/or RECIST 1.1 (as assessed by the investigator and confirmed by BIRC), withdrawal of consent, pregnancy, lost to follow-up, or death.

For all participants, treatment with capmatinib may be continued beyond initial progression disease (PD) as per RANO-BM criteria and/or RECIST 1.1 (as assessed by the investigator and confirmed by BIRC) if, in the judgment of the investigator, there is evidence of clinical benefit, and the participant wishes to continue on the study treatment.

After treatment discontinuation, all participants will be followed for safety evaluations during the safety follow-up period, and the participant's status will be collected every 12 weeks as part of the survival follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed stage IV (according to Version 8 of the American Joint Committee on Cancer (AJCC)) NSCLC that is EGFR wt, ALK rearrangement negative as assessed by a validated test as part of the participant's standard of care and has MET∆ex14 mutation per Novartis-designated central laboratory or (US only) locally with FoundationOne Companion Diagnostic (F1CDx) .
* Treatment naïve or up to two prior lines of systemic therapy for stage IIIb-IV NSCLC
* Measurable intracranial lesions:

  1. Cohort 1 and Cohort 2 (without leptomeningeal carcinoma): At least 1 measurable intracranial lesion per RANO-BM criteria, documented by a radiologist/neuroradiologist (treated or untreated).
  2. Cohort 2 (with leptomeningeal carcinoma): participants with leptomeningeal carcinoma may not have measurable lesions. In this circumstance, the participant's disease will be considered to have non-target lesions only at baseline and their response based on descriptive clinical criteria by physician assessment.
* Capable of undergoing magnetic resonance imaging (MRI)
* ECOG performance status of 0 or 1

Exclusion Criteria:

* Only for Cohort 1: any neurological symptoms related to brain metastases
* For participants in Cohort 2 with prior brain therapy: Treatment with stereotactic radiosurgery within 14 days prior to the start of study treatment or treatment with WBRT within 14 days prior to the start of study treatment
* Prior treatment with any MET targeting therapy or HGF inhibitor
* Participants with other known druggable molecular alterations (such as ROS1 translocation or BRAF mutation) who might be candidates to alternative targeted therapies as applicable per local regulations and treatment guidelines
* Presence or history of ILD or interstitial pneumonitis, including clinically significant radiation pneumonitis (i.e., affecting activities of daily living or requiring therapeutic intervention)
* Clinically significant, uncontrolled heart diseases including History of familial long QT syndrome, sudden death or congenital long QT syndrome

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-11-11 (Estimated); Primary Completion 2023-11-17 (Estimated); Study Completion 2023-11-17 (Estimated)

PRIMARY OUTCOMES:
Overall Intracranial Response Rate (OIRR) in Cohort 1 by Blinded Independent Review Committee (BIRC) review | Up to 36 months
  Overall Intracranial Response Rate (OIRR) in Cohort 1, defined as the proportion of participants with a confirmed best intracranial overall response of Complete Response (CR) or Partial Response (PR) per RANO-BM criteria as assessed by BIRC review

SECONDARY OUTCOMES:
Overall Intracranial Response Rate (OIRR) in Cohort 1 by investigator review | Up to 36 months
  Overall Intracranial Response Rate (OIRR) in Cohort 1, defined as the proportion of participants with a confirmed best intracranial overall response of Complete Response (CR) or Partial Response (PR) per RANO-BM criteria as assessed by investigator review
Intracranial Disease Control Rate (IDCR) by investigator and BIRC review | Up to 36 months
  Intracranial Disease Control Rate (IDCR) per RANO-BM criteria as assessed by investigator review and by BIRC review
Time to intracranial tumor Response (TTIR) by investigator and BIRC review | Up to 36 months
  Time to intracranial tumor Response (TTIR) per RANO-BM criteria as assessed by investigator review and by BIRC review
Duration of Intracranial Response (DOIR) by investigator and BIRC review | Up to 36 months
  Duration of Intracranial Response (DOIR) per RANO-BM as assessed by investigator review and by BIRC review
Overall Intracranial Response Rate (OIRR) in Cohort 2 by investigator and BIRC review | Up to 36 months
  Overall Intracranial Response Rate (OIRR) per RANO-BM criteria in Cohort 2 by investigator review and by BIRC review
Overall Extracranial Response Rate (OERR) by investigator and BIRC review | Up to 36 months
  Overall Extracranial Response Rate (OERR) per RECIST 1.1 by investigator review and by BIRC review
Extracranial Disease Control Rate (EDCR) by investigator and BIRC review | Up to 36 months
  Extracranial Disease Control Rate (EDCR) per RECIST 1.1 by investigator and BIRC review
Time to Extracranial Response (TTER) by investigator and BIRC review | Up to 36 months
  Time to Extracranial Response (TTER) per RECIST 1.1 by investigator review and by BIRC review
Duration of Extracranial Response (DOER) by investigator and BIRC review | Up to 36 months
  Duration of Extracranial Response (DOER) per RECIST 1.1 by investigator review and by BIRC review
Overall Response Rate (ORR) per RECIST 1.1 by investigator and BIRC review | Up to 36 months
  Overall Response Rate (ORR) in the whole body per RECIST 1.1 by investigator review and by BIRC review
Time to response (TTR) by investigator and BIRC review | Up to 36 months
  Time to response (TTR) in the whole body per RECIST 1.1 by investigator review and by BIRC review
Duration of response (DOR) by investigator and BIRC review | Up to 36 months
  Duration of response (DOR) in the whole body per RECIST 1.1 by investigator review and by BIRC review
Progression free survival (PFS) by investigator and BIRC review | Up to 36 months
  Progression free survival (PFS) in the whole body per RECIST 1.1 by investigator review and by BIRC review
Overall survival (OS) | Up to 36 months
  Overall survival (OS) is defined as the time from the date of start of treatment to the date of death due to any cause.
Percentage of patients with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 36 months
  Safety profile of capmatinib. Incidence and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) including any clinically significant lab, vital signs, ECG abnormalities that are captured as an AE
Number of participants with dose interruptions | Up to 29 months
  Tolerability measured by the number of subjects who have interruptions of study treatment
Number of participants with dose reductions | Up to 29 months
  Tolerability measured by the number of subjects who have reductions of study treatment
Dose intensity | Up to 29 months
  Tolerability measured by the dose intensity of study drug computed as the ratio of actual cumulative dose received and actual duration of exposure
Time to deterioration in Functional Assessment of Cancer Therapy (FACT)-Brain Symptom Index (FBrSI) scores in Cohort 1 | Day 1 and 15 of Cycle 1, Day 1 of cycles 2 to 11 and then every other cycle until end of treatment (up to 29 months). Cycle=28 days
  Time to deterioration in symptoms of brain metastases in Cohort 1 with the Functional Assessment of Cancer Therapy (FACT)-Brain Symptom Index (FBrSI) (a standardized questionnaire developed to assess the quality of life of cancer patients)
Change from baseline in score as per FACT-Brain Symptom Index (FBrSI) in Cohort 2 | Day 1 and 15 of Cycle 1, Day 1 of cycles 2 to 11 and then every other cycle until end of treatment (up to 29 months). Cycle=28 days
  Change from baseline in symptoms of brain metastases in Cohort 2 with the FACT-Brain Symptom Index (FBrSI) (a standardized questionnaire developed to assess the quality of life of cancer patients)
Change from baseline in score as per European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-C30 | Day 1 of cycle 1 to 11 and then every other cycle until end of treatment (up to 29 months). Cycle=28 days
  Change from baseline in lung cancer related symptoms, functioning and other domains of HRQoL in both cohorts with the EORTC QLQ-C30 (a 30-item questionnaire developed to assess the quality of life of cancer patients)
Change from baseline in score as per European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Lung Cancer Module (QLQ-LC13) | Day 1 of cycle 1 to 11 and then every other cycle until end of treatment (up to 29 months). Cycle=28 days
  Change from baseline in lung cancer related symptoms, functioning and other domains of HRQoL in both cohorts with the QLQ-LC13 (a 13-item questionnaire developed to assess the quality of life of cancer patients)
Change from baseline in score as per European Quality of Life 5-Dimension 5-Level (EQ-5D-5L) questionnaire | Day 1 of cycle 1 to 11 and then every other cycle until end of treatment (up to 29 months). Cycle=28 days
  Change from baseline in lung cancer related symptoms, functioning and other domains of HRQoL in both cohorts with the EQ-5D-5L (a standardized questionnaire developed to assess the quality of life of cancer patients)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com